CLINICAL TRIAL: NCT00044343
Title: An Open-Label, Multicenter, Phase II Study of Oral Lapatinib (GW572016) as Single Agent, Second-Line Therapy in Subjects With Metastatic Colorectal Cancer Who Have Progressed on First-Line Therapy With 5-Fluorouracil in Combination With Irinotecan or Oxaliplatin
Brief Title: GW572016, An Oral Drug For Colorectal Cancer Patients Having Prior Therapy With 5-FU Plus CPT-11 And/Or Oxaliplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF20004
Record Dates: First submitted 2002-08-26; First posted 2002-08-28 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; EGFR inhibitor; lapatinib; metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Lapatinib

INTERVENTIONS:
Drug: lapatinib

SUMMARY:
The purpose of this study is to determine the efficacy of an oral investigational drug in patients with refractory metastatic colorectal cancer after receiving prior therapy with 5-fluorouracil in combination with irinotecan and/or oxaliplatin.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed informed consent.
* Refractory Stage IV metastatic colorectal cancer.
* Received at least 2 cycles of first-line therapy with intravenous 5-FU (5-fluorouracil) in combination with CPT-11 (irinotecan) and/or oxaliplatin.
* No more than one prior therapy.
* Tumor tissue available for testing.
* 4 weeks since first-line cancer regimen.
* Able to swallow and retain oral medication.
* Cardiac ejection fraction within the institutional range of normal as measured by MUGA (Multiple Gated Acquisition Scan).
* Adequate kidney and liver function.
* Adequate bone marrow function.

Exclusion Criteria:

* Pregnant or lactating female.
* Conditions that would affect absorption of an oral drug
* First-line regimen did not include 5-fluorouracil with irinotecan and/or oxaliplatin.
* Serious medical or psychiatric disorder that would interfere with the patient''s safety or informed consent.
* Severe cardiovascular disease or cardiac (heart) disease requiring a device.
* Active infection.
* Brain metastases.
* Concurrent cancer therapy or investigational therapy.
* Use of oral or intravenous steroids.
* Unresolved or unstable, serious toxicity from prior therapy.
* Prior therapy with an EGFR (Endothelial Growth Factor Receptor) and/or erbB-2 inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2002-09; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Tumor response rate (complete or partial). | 6 Months

SECONDARY OUTCOMES:
Time to response duration of response time to progression 4-month progression-free survival 6-month progression-free survival overall survival safety data biomarkers | 6 Month

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trial, MD, Study Director — GlaxoSmithKline
Locations (56):
- United States (49):
  - GSK Clinical Trials Call Center, Los Angeles, California
  - GSK Clinical Trials Call Center, Poway, California
  - GSK Clinical Trials Call Center, Torrington, Connecticut
  - GSK Clinical Trials Call Center, Boca Raton, Florida
  - GSK Clinical Trials Call Center, Fort Lauderdale, Florida
  - GSK Clinical Trials Call Center, Fort Myers, Florida
  - GSK Clinical Trials Call Center, Miami, Florida
  - GSK Clinical Trials Call Center, Sarasota, Florida
  - GSK Clinical Trials Call Center, Atlanta, Georgia
  - GSK Clinical Trials Call Center, Marietta, Georgia
  - GSK Clinical Trials Call Center, Terre Haute, Indiana
  - GSK Clinical Trials Call Center, Des Moines, Iowa
  - GSK Clinical Trials Call Center, Lafayette, Louisiana
  - GSK Clinical Trials Call Center, New Orleans, Louisiana
  - GSK Clinical Trials Call Center, Rockville, Maryland
  - GSK Clinical Trials Call Center, Wellesley, Massachusetts
  - GSK Clinical Trials Call Center, Saint Charles, Missouri
  - GSK Clinical Trials Call Center, Saint Joseph, Missouri
  - GSK Clinical Trials Call Center, St Louis, Missouri
  - GSK Clinical Trials Call Center, Billings, Montana
  - GSK Clinical Trials Call Center, Great Falls, Montana
  - GSK Clinical Trials Call Center, Omaha, Nebraska
  - GSK Clinical Trials Call Center, Hooksett, New Hampshire
  - GSK Clinical Trials Call Center, Morristown, New Jersey
  - GSK Clinical Trials Call Center, Summit, New Jersey
  - GSK Clinical Trials Call Center, Armonk, New York
  - GSK Clinical Trials Call Center, Brooklyn, New York
  - GSK Clinical Trials Call Center, New York, New York
  - GSK Clinical Trials Call Center, Rockville Centre, New York
  - GSK Clinical Trials Call Center, White Plains, New York
  - GSK Clinical Trials Call Center, Charlotte, North Carolina
  - GSK Clinical Trials Call Center, Goldsboro, North Carolina
  - GSK Clinical Trials Call Center, Greensboro, North Carolina
  - GSK Clinical Trials Call Center, Greenville, North Carolina
  - GSK Clinical Trials Call Center, Hickory, North Carolina
  - GSK Clinical Trials Call Center, Cincinnati, Ohio
  - GSK Clinical Trials Call Center, Altoona, Pennsylvania
  - GSK Clinical Trials Call Center, Bethlehem, Pennsylvania
  - GSK Clinical Trials Call Center, Hershey, Pennsylvania
  - GSK Clinical Trials Call Center, Kingston, Pennsylvania
  - GSK Clinical Trials Call Center, Lancaster, Pennsylvania
  - GSK Clinical Trials Call Center, Spartanburg, South Carolina
  - GSK Clinical Trials Call Center, West Columbia, South Carolina
  - GSK Clinical Trials Call Center, Germantown, Tennessee
  - GSK Clinical Trials Call Center, Nashville, Tennessee
  - GSK Clinical Trials Call Center, Burien, Washington
  - GSK Clinical Trials Call Center, Olympia, Washington
  - GSK Clinical Trials Call Center, Puyallup, Washington
  - GSK Clinical Trials Call Center, Yakima, Washington
- Canada (7):
  - GSK Clinical Trials Call Center, Edmonton, Alberta
  - GSK Clinical Trials Call Center, Winnipeg, Manitoba
  - GSK Clinical Trials Call Center, Greater Sudbury, Ontario
  - GSK Clinical Trials Call Center, Thunder Bay, Ontario
  - GSK Clinical Trials Call Center, Lévis, Quebec
  - GSK Clinical Trials Call Center, Montreal, Quebec
  - GSK Clinical Trials Call Center, Sainte-Foy, Quebec